CLINICAL TRIAL: NCT02197819
Title: A Randomized Evaluation of Emergent Immobilization in External Rotation in the Management of Acute Anterior Dislocations of the Shoulder
Acronym: EERAADS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow patient enrolment
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EERAADS
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2018-04

CONDITIONS: Primary Anterior Shoulder Dislocation
MeSH Terms: interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Rotation Brace (Experimental): Shoulder placed in an external rotation brace for 4 weeks
  Interventions: Device: External Rotation Brace
- Traditional Sling (Active Comparator): Patient placed in traditional sling
  Interventions: Device: Sling

INTERVENTIONS:
Device: Sling
  Arms: Traditional Sling
Device: External Rotation Brace
  Arms: External Rotation Brace

SUMMARY:
Shoulder dislocations are quite common, the prevalence over a lifetime being estimated at 2% in the general population. In young patients, recurrence after a primary dislocation is also common (~60%) and multiple recurrent episodes can cause significant disability over time. Following initial reduction of the joint, the traditional treatment for primary shoulder dislocations has been immobilization in a sling, with the arm in a position of adduction and internal rotation. The length of the immobilization period is controversial, however most authors would recommend between three to six weeks in a sling followed by several months of rehabilitation to include range of motion and strengthening exercises. The clinical course of patients after this approach has been extensively investigated. Of particular interest is the relatively high rate of recurrent instability in young patients, reported to be between 17 and 96%.

A prospective randomized trial is needed to determine whether in young patients (16-30 yrs of age) following reduction of a first-time traumatic anterior shoulder dislocation, does EMERGENT (<4 hours post reduction) immobilization of the affected shoulder in external rotation reduce the rate of recurrent instability experienced within 12 months versus emergent immobilization in a traditional internal rotation sling? Eligible patients will be randomly allocated to the sling or ER brace. The results of this study will provide the best evidence for choosing emergent immobilization for shoulder dislocations.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients between 18 - 35 years of age inclusive
* Patient is seen within 24 hours from time of injury.
* Sustained an acute, first-time, traumatic anterior dislocation of the shoulder as defined by;
* Mechanism of abduction, external rotation
* Sudden pain in the shoulder
* Manipulative reduction required or
* Radiograph documenting a dislocated joint
* Willing to participate in follow-up for at least 24 months.

Exclusion Criteria:

* Incompetent or unwilling to consent
* Inability or unwillingness to comply with rehabilitative protocol or required follow-up assessments.
* Previous instability of the affected shoulder
* Significant associated fracture (Exception Hill Sachs or bankart lesions)
* Concomitant ipsilateral upper extremity injuries which may affect the patient's ability to participate in, or benefit from, a rehabilitative program.
* Neurovascular compromise of the affected limb
* A medical condition making the patient unable to wear a brace or sling
* Patient is seen within 24 hours from time of injury

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Re-dislocation of shoulder | within 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada